CLINICAL TRIAL: NCT05392361
Title: Effect of Baclofen Treatment on Nocturnal Muscle Cramps in Patients With Lumbar Spinal Stenosis: a Randomized Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4-2022-0360
Record Dates: First submitted 2022-05-18; First posted 2022-05-26 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Lumbar Spinal Stenosis With Nocturnal Calf Cramps
Keywords: baclofen; spinal stenosis; nocturnal calf cramps
MeSH Terms: conditions — Spinal Stenosis | interventions — Gabapentin; Therapeutics; Baclofen

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Active Comparator): conservative management for spinal stenosis
  Interventions: Drug: gabapentin (neurontin® capsule 300mg) treatment
- baclofen group (Experimental): conservative management for spinal stenosis plus baclofen treatment
  Interventions: Drug: baclofen (baclofen Tab. 10mg) treatment

INTERVENTIONS:
Drug: gabapentin (neurontin® capsule 300mg) treatment — Taking gabapentin (neurontin® capsule 300mg, Pfizer) medication at night as a conservative treatment
  Arms: control group
Drug: baclofen (baclofen Tab. 10mg) treatment — Taking baclofen (baclofen Tab. 10mg, Handok co, Seoul, Korea) medication at night.
  Arms: baclofen group

SUMMARY:
Nocturnal calf cramps is a common complaint in patients with lumbar spinal stenosis. The purpose of this study is to evaluate the effect of baclofen in lumbar spinal stenosis patients receiving conservative therapy. We will compare pain score, insomnia severity, functional ability and patient satisfaction between control (conservative management for spinal stenosis) and baclofen group (conservative management for spinal stenosis plus baclofen treatment).

ELIGIBILITY:
Inclusion Criteria:

1. diagnosed lumbar spinal stenosis with MRI finding
2. nocturnal calf cramps symptoms at least once per week

Exclusion Criteria:

1. electrolyte disorder
2. congenital muscle disease
3. muscle cramps related medication (statins, diuretics, calcium channel blockers, anticonvulsants etc.)
4. cognitive impairments

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-06-09 (Actual); Primary Completion 2023-03-24 (Actual); Study Completion 2023-03-24 (Actual)

PRIMARY OUTCOMES:
Pain score | follow up 4 weeks
  A comparison of pain score between control (conservative management for spinal stenosis) and baclofen group (conservative management for spinal stenosis plus baclofen treatment).
  The pain score will be measured using NRS (Numeric Rating Scale) on a scale from 0-10, with 0 representing "no pain" and 10 "worst possible pain".

SECONDARY OUTCOMES:
Frequency and severity of nocturnal calf cramps | follow up 4 weeks, 12 weeks
  The frequency(number) and the severity of nocturnal calf cramps that occurred in a week before each time frame will be investigated. The severity of nocturnal calf cramps will be measured by 0-4 point scale (0, no pain; 1, mild pain that disappeared immediately and tolerable; 2, moderate pain accompanied by pain enough to wake up from sleep; 3, severe pain accompanied by pain enough to wake up from sleep for a long time; 4, severe pain that lasted for a long time and affected a daily life of the next day)
Insomnia severity index | follow up 4 weeks, 12 weeks
Oswestry Disability Index | follow up 4 weeks, 12 weeks
Patient satisfaction (PGIC) | follow up 4 weeks, 12 weeks
  Patient satisfaction with treatment at 12 weeks after treatment will be measured by 7-point Patient Global Impression of Change (PGIC; 1, very much improved; 2, much improved; 3, minimally improved; 4, no change; 5, minimally worse; 6, much worse; 7, very much worse)

CONTACTS AND LOCATIONS:
Overall Officials: Shin Hyung Kim, Principal Investigator — Anesthesiology and Pain Medicine, Yonsei University College of Medicine
Locations (1):
- Yonsei University Health System, Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim HJ, Yoon KB, Kang M, Lee HW, Kim SH. Use of Baclofen as a Treatment for Nocturnal Calf Cramps in Individuals With Lumbar Spinal Stenosis: A Prospective Randomized Study. Am J Phys Med Rehabil. 2024 May 1;103(5):384-389. doi: 10.1097/PHM.0000000000002364. Epub 2023 Nov 22. PMID 38063320